CLINICAL TRIAL: NCT06281015
Title: Ultra-Fast Whole-Body Bone Tomoscintigraphies Achieved With a High-Sensitivity 360° CZT Camera and a Dedicated Deep Learning Noise Reduction Algorithm
Brief Title: Artificial Intelligence and Bone Tomoscintigraphies Achieved With CZT Camera
Acronym: IATOS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Achraf BAHLOUL, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI095-407
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bone Lesion
MeSH Terms: interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Whole-body bone single photon emission tomography (SPECT) for detection or follow-up of bone metastasis — Cancer patients referred to fast whole-body bone for detection or follow-up of bone metastasis were retrospectively included in this study.

SUMMARY:
This study aimed to determine whether the whole-body bone Single Photon Emission Computed Tomography (SPECT) recording times of around 10 minutes, routinely provided by a high-sensitivity 360 degrees cadmium and zinc telluride (CZT) camera, can be further reduced by a deep learning noise reduction (DLNR) algorithm.

DETAILED DESCRIPTION:
This study aimed to determine the extent to which fast whole-body bone-SPECT recording times, routinely obtained with a high-sensitivity 360 degrees CZT-camera and rather low injected activities, can be further reduced using the DLNR algorithm.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to fast whole-body bone single photon emission tomography for detection or follow-up of bone metastasis

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nineteen cancer patients (8 women, 11 men) referred to fast whole-body bone single photon emission tomography for detection or follow-up of bone metastasis were retrospectively included in this study.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Assess a dedicated deep learning noise reduction algorithm | one day
  A deep learning noise reduction algorithm was applied on whole-body images recorded

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France